CLINICAL TRIAL: NCT04452513
Title: A Prospective Clinical Study of Phenylketonuria (PKU)
Status: Completed | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 307-902
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2022-09

CONDITIONS: Phenylketonurias
Keywords: PKU; Phenylketonuria; PAH Deficiency
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a study for adults and children ≥ 14 years old who have Phenylketonuria (PKU) with uncontrolled plasma Phe levels. No clinical intervention or study drug is provided by BioMarin in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with diagnosis of PKU which is a condition characterized by PAH deficiency
* Ability and willingness to maintain dietary protein intake consistent with baseline intake
* Willingness and capable per investigator opinion to comply with study procedures and requirements
* Plasma Phe Levels > 600umol/L

Exclusion Criteria:

* Clinically significant liver dysfunction or disease
* Prior treatment with gene therapy
* Any condition that, in the opinion of the investigator or Sponsor, would prevent the subject from fully complying with the requirements of the study

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PKU Patients 14 years or older with uncontrolled plasma Phe levels
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Change in Plasma Phe Levels | through study completion, an average of 2 years

SECONDARY OUTCOMES:
Change in dietary protein intake from medical and intact food | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Children's Hosptial of Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Ann & Robert H. Lurie Chilren's Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Boston Children's Hospital, Boston, Massachusetts
  - Morristown Medical Center, Morristown, New Jersey
  - Oregon Health & Science University, Portland, Oregon
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Clinic for Special Children, Strasburg, Pennsylvania
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Medical College of Wisconsin, Wauwatosa, Wisconsin